CLINICAL TRIAL: NCT03712371
Title: Phase 1b/2 Study of Chitosan for Pharmacologic Manipulation of AGE (Advanced Glycation Endproducts) Levels in Prostate Cancer Patients
Brief Title: Study of Chitosan for Pharmacologic Manipulation of AGE Levels in Prostate Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim study results were not favorable to continue with further enrollment.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 102928
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Results first posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Chitosan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chitosan Dose Escalation (Experimental): The starting dose for Chitosan is 500mg twice daily, the second dose level is 1000mg twice daily, the third dose level is 1500mg twice daily and the fourth dose level is 2000mg twice daily. Safety evaluation is 28 days in length and total dose administration is 85 days in length.
  Interventions: Drug: Chitosan

INTERVENTIONS:
Drug: Chitosan — Increasing dose levels from 500mg twice daily to 2000mg twice daily for up to 85 days.

SUMMARY:
This study will examine the utility of chitosan for reduction of blood or tissue levels of AGEs in patients with prostate cancer who are clinically stable on androgen-deprivation therapy.

DETAILED DESCRIPTION:
The overall goal of this study is to identify a safe dose of the metabolic supplement, Chitosan that can help reduce AGE (advanced glycation endproducts) levels in patients with prostate cancer. Chitosan is a naturally occurring substance found in shellfish. This study will be using Chitosan prepared from the shells of cold-water shrimp. Chitosan is approved by the FDA for use in wound dressings and has been used in published clinical trials for weight loss but is not approved for the purposes of this study. AGEs are a type of metabolite, or substance, found in food and produced in the body. The researchers helping conduct this study have found a potential link between AGE levels and cancer. Participation in this study will require three study visits over the course of about 3 months. During these visits subjects will be asked to provide blood and stool samples as well as complete surveys about their quality of life.

ELIGIBILITY:
Inclusion:

1. Confirmation of adenocarcinoma of the prostate that is documented by one of the following: pathology report or clinic note with documented history of prostate cancer.
2. Subjects must be receiving ADT with a GnRH agonist or antagonist, with or without an anti-androgen or testosterone synthesis inhibitor. The current testosterone level must be documented to be <50ng/dL at enrollment. Subjects whose ADT is interrupted may enroll or continue on study as long as the testosterone is documented to remain <50ng/dL for the entire duration of study participation. Subjects who have undergone orchiectomy are also eligible.
3. Subjects must have adequate hematologic, renal, and hepatic function at baseline, as follows:

   * Hematology parameters: ANC >1000/mcL, platelets > 100,000/mcL, Hgb >8.0gm/dL
   * Renal Function: eGFR of ≥ 45mls/min using Cockgroft and Gault formula
   * Liver Function: Total bilirubin ≤ULN, AST and ALT <1.5x ULN
4. Able to swallow and retain oral medication
5. ECOG performance status of 0 - 2
6. Ability to sign written informed consent
7. Testosterone level <50ng/dL at time of enrollment.
8. Age 18 or older.
9. May have had prior radiation therapy, surgery, or cryoablation for primary prostate cancer
10. May have had prior cytotoxic chemotherapy for metastatic prostate cancer, prior treatment with genomically-targeted agents, or Provenge

Exclusion:

1. Known allergy to chitosan or shellfish.
2. History of receiving more than 2 classes of ADT.
3. Chronic constipation (BM < 3x weekly), history of malabsorption or history of daily laxative use.
4. Patients requiring medication administration with lunch or dinner or at a frequency of three or more times per day are not eligible.
5. Current use of chitosan, sevelamer, and/or glucosamine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lilly, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Chitosan 500mg twice daily for a 28-day DLT evaluation period, and for a total treatment duration of 85 days.
- Dose Level 2: Chitosan 1000mg twice daily for a 28-day DLT evaluation period, and for a total treatment duration of 85 days.
- Dose Level 3: Chitosan 1500mg twice daily for a 28-day DLT evaluation period, and for a total treatment duration of 85 days.
- Dose Level 4: Chitosan 2000mg twice daily for a 28-day DLT evaluation period, and for a total treatment duration of 85 days.
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 2
Not Completed | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Four dose levels of Chitosan twice daily for a 28-day DLT evaluation period, and continuing for a total treatment duration of 85 days.
  Dose level 1: 500mg, Dose level 2: 1000mg, Dose level 3: 1500mg, Dose level 4: 2000mg.
Groups:
- Chitosan Dose Level 1: ChChitosan dosing 500mg orally twice daily for 85 days.
- Chitosan Dose Level 2: Chitosan dosing 1000mg orally twice daily for 85 days.
- Chitosan Dose Level 3: Chitosan dosing 1500mg orally twice daily for 85 days.
- Chitosan Dose Level 4: Chitosan dosing 2000mg orally twice daily for 85 days.
- Total: Total of all reporting groups
Arm/Group | Chitosan Dose Level 1 | Chitosan Dose Level 2 | Chitosan Dose Level 3 | Chitosan Dose Level 4 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 1 | 1
  >=65 years | 3 | 3 | 3 | 2 | 11
Age, Continuous [Median (Full Range); unit: years] | 68 [66 to 70] | 75 [68 to 83] | 73 [69 to 75] | 69 [61 to 74] | 69.5 [61 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 3 | 2 | 3 | 3 | 11
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose as Assessed by Number of Participants Who Experienced a Dose Limiting Toxicity
Description: The maximum tolerated dose is defined as the dose that produces no more than 1 dose-limiting toxicity (DLT)in 6 subjects. Per protocol a DLT is defined as Grade 3 or higher hypophosphatemia and/ or Grade 3 or higher of any of the following toxicities, that the investigator deems related to chitosan, that do not improve or resolve within 7 days of onset: flatulence, increased stool bulkiness, bloating, nausea, heartburn
Time Frame: 112 days
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Redox Status (RedoxSys, Serum Oxidized Glutathione)
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Inflammation (Plasma Cytokines, Toll-like Receptor Signaling)
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Insulin Resistance (HOMA-IR)
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Changes in Bowel Permeability (Plasma Endotoxin)
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Changes in Microbiome Diversity (16s rDNA Sequencing)
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Correlate Changes in Serum AGE Levels (Pan-AGE, Carboxymethyllysine, Methylglyoxal
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Measure the Frequency of a > 30% Reduction in Total AGE Levels From the Pretreatment Level.
Description: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Time Frame: 112 days
Population: No participants were analyzed for this outcome, therefore no data was collected. Study was terminated.
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 5 months, 14 days
Description: NCI CTCAE version 5.0
Groups:
- Chitosan Dose Level 1: Chitosan 500mg orally twice daily for a 28 day DLT period and for a total dosing regimen of 85 days.
- Chitosan Dose Level 2: Chitosan 1000mg orally twice daily for a 28 day DLT period and for a total dosing regimen of 85 days.
- Chitosan Dose Level 3: Chitosan 1500mg orally twice daily for a 28 day DLT period and for a total dosing regimen of 85 days.
- Chitosan Dose Level 4: Chitosan 2000mg orally twice daily for a 28 day DLT period and for a total dosing regimen of 85 days.
Arm/Group | Chitosan Dose Level 1 | Chitosan Dose Level 2 | Chitosan Dose Level 3 | Chitosan Dose Level 4
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chitosan Dose Level 1 (N=3) | Chitosan Dose Level 2 (N=3) | Chitosan Dose Level 3 (N=3) | Chitosan Dose Level 4 (N=3)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chitosan Dose Level 1 (N=3) | Chitosan Dose Level 2 (N=3) | Chitosan Dose Level 3 (N=3) | Chitosan Dose Level 4 (N=3)
dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
lightheadedness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
dry mouth (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
bladder neck contracture (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypersomnia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
frequent urination (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
increased stool bulkiness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
difficulty with balance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cognitive slowness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
decreased muscle mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
increased urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
neuropathic pain - limbs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
eye redness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
blurred vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
generalized discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to analysis of AGE assay blood specimens demonstrating a lack of efficacy with the test article. Due to early termination, none of the secondary outcomes were measured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT03712371/Prot_SAP_000.pdf